CLINICAL TRIAL: NCT02276651
Title: A Prospective Multicenter Observational Trial of a Therapeutic Platelet Transfusion Regimen for Patients With Acute Myeloid Leukemia in Consolidation Chemotherapy
Brief Title: Observational Trial of a Therapeutic Platelet Transfusion Regimen
Status: Terminated | Type: Observational
Why Stopped: Insufficient recruitment
Sponsor: Klinikum Nürnberg (Other)
Collaborators: Technische Universität Dresden (Other); University Hospital Heidelberg (Other); Klinikum Chemnitz gGmbH (Other); University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Dr Kerstin Schäfer-Eckart, Principal Investigator, Klinikum Nürnberg
Other Study IDs: 001
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Acute Myeloid Leukemia; Thrombocytopenia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Application of a therapeutic platelet transfusion Regimen in patients with acute myeloid leukemia in complete Remission (consolidation therapy)

DETAILED DESCRIPTION:
For the participants a therapeutic regimen for platelet transfusions will be applied: for clinically stable patients platelet Transfusion will be given in case of bleeding WHO II° or higher, for clinically instable patients platelet transfusion will be given at the decretion of the attending physician.

Patients with sepsis, septic shock or infections with Infiltration of organs (e.g. invasive aspergillosis), plasmatic coagulation disorders or sudden or increasing headache with or without neurologic symptoms should receive prophylactic platelet Transfusion, if their platelet Count is less then 10/nl. Otherwise no prophylactic platelet Transfusion will be given irrespective of the actual platelet Count.

As Primary study endpoint The incidence of bleeding episodes WHO grade III an IV will be documented. The bleeding incidence will then be compared to a historic cohort.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia in complete remission

Exclusion Criteria:

* plasmatic coagulopathy
* history of severe bleeding complications in chemotherapy induced thrombocytopenia
* no increment in platelets after platelet transfusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with acute myeloid leukemia in complete remission receiving postremission chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
Bleeding Grade III and IV (WHO) | Patients will be followed for the phase of thrombocytopenia after chemotherapy, an expected average of about 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Schaefer-Eckart, MD, Principal Investigator — Klinikum Nürnberg
Locations (1):
- Klinikum Nurnberg, Nuremberg, Germany

REFERENCES:
- [Background] Wandt H, Schaefer-Eckart K, Wendelin K, Pilz B, Wilhelm M, Thalheimer M, Mahlknecht U, Ho A, Schaich M, Kramer M, Kaufmann M, Leimer L, Schwerdtfeger R, Conradi R, Dolken G, Klenner A, Hanel M, Herbst R, Junghanss C, Ehninger G; Study Alliance Leukemia. Therapeutic platelet transfusion versus routine prophylactic transfusion in patients with haematological malignancies: an open-label, multicentre, randomised study. Lancet. 2012 Oct 13;380(9850):1309-16. doi: 10.1016/S0140-6736(12)60689-8. Epub 2012 Aug 8. PMID 22877506
- [Background] Wandt H, Schafer-Eckart K, Ehninger G. Prophylactic platelet transfusion. N Engl J Med. 2013 Aug 8;369(6):577. doi: 10.1056/NEJMc1307163. No abstract available. PMID 23924012
- [Background] Wandt H, Schaefer-Eckart K, Frank M, Birkmann J, Wilhelm M. A therapeutic platelet transfusion strategy is safe and feasible in patients after autologous peripheral blood stem cell transplantation. Bone Marrow Transplant. 2006 Feb;37(4):387-92. doi: 10.1038/sj.bmt.1705246. PMID 16400342
- [Background] Wandt H, Frank M, Ehninger G, Schneider C, Brack N, Daoud A, Fackler-Schwalbe I, Fischer J, Gackle R, Geer T, Harms P, Loffler B, Ohl S, Otremba B, Raab M, Schonrock-Nabulsi P, Strobel G, Winter R, Link H. Safety and cost effectiveness of a 10 x 10(9)/L trigger for prophylactic platelet transfusions compared with the traditional 20 x 10(9)/L trigger: a prospective comparative trial in 105 patients with acute myeloid leukemia. Blood. 1998 May 15;91(10):3601-6. PMID 9572994
- [Background] Wandt H, Ehninger G, Gallmeier WM. New strategies for prophylactic platelet transfusion in patients with hematologic diseases. Oncologist. 2001;6(5):446-50. doi: 10.1634/theoncologist.6-5-446. PMID 11675523